CLINICAL TRIAL: NCT00786032
Title: Cooperative Studies Program (CSP) #567 - A Clinical Demonstration of EEG Brain-computer Interface for ALS Patients
Brief Title: A Clinical Demonstration of EEG Brain-computer Interface for ALS Patients
Acronym: ALS
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 567
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Amyotrophic Lateral Sclerosis; Brain Computer Interface (BCI); Lou Gehrig's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BCI Device: All participants will use the BCI System as a means of communication.
  Interventions: Device: BCI Device

INTERVENTIONS:
Device: BCI Device — A Brain Computer interface or BCI records brain signals and analyzes them to derive device commands. BCIs give their users communication and control channels that do not depend on peripheral nerves and muscles.
  Other Names: Brain Computer Interface Device (BCI)

SUMMARY:
The goal of this VA demonstration project is to show that the Brain-computer interface (BCI) technology is a clinically practical and important new communication and control option that can improve the lives of veterans with amyotrophic lateral sclerosis (ALS). The project will test four well-supported hypotheses: (1) that people with ALS who find (or will soon find) conventional assistive technology inadequate can and will use a BCI system for important purposes in their daily lives without close technical oversight, 2) they will continue and even increase this use throughout the period of the study, (3) that BCI use will improve their lives, and 4) BCI will improve the lives of their families and caregivers.

DETAILED DESCRIPTION:
People affected by severe motor disorders such as amyotrophic lateral sclerosis (ALS) need alternative methods for communication and control. They may not be able to use even the most basic conventional assistive technologies, which all rely in one way or another on muscles. For these people, communication and control technology that does not depend on neuromuscular function is essential. Brain-computer interfaces (BCIs) can give these individuals communication and control capacity that does not depend on nerves and muscles. It has been shown that even people who are almost completely paralyzed can control sensor motor rhythms and other features of scalp-recorded electroencephalographic (EEG) activity and that they can use this control to move a computer cursor in one or two dimensions, to select letters or icons, or even to move a robotic arm. The group is now focused on developing clinically practical BCI applications, translating them from the laboratory into people's homes, and establishing that they can have a positive impact on the lives of people with severe disabilities.

The goal of this VA demonstration project is to show that BCI technology is a clinically practical and important new communication and control option that can improve the lives of veterans with amyotrophic lateral sclerosis (ALS). The project will test four well-supported hypotheses: (1) that people with ALS who find (or will soon find) conventional assistive technology inadequate can and will use a BCI system for important purposes in their daily lives without close technical oversight, 2) they will continue and even increase this use throughout the period of the study, (3) that BCI use will improve their lives, and 4) BCI will improve the lives of their families and caregivers.

In accord with these hypotheses, the aims are:

Aim 1: To recruit 2-4 person teams of VA health professionals (e.g., physicians, nurses, nurse- practitioners, physician's assistants, EEG technicians, therapists, rehabilitation specialists, medical researchers) at each of 5-6 participating VA centers, and train them in the use and ongoing support of the BCI home system. These teams will use the VA ALS database, local ALS Association affiliates, and VA clinics to identify and recruit at each site 3-4 patients with ALS who are not adequately served by conventional assistive technology; have stable physical and social environments; and have caregivers with basic computer skills who are willing to support BCI use. The VA teams will set up BCI systems in the patients' homes and teach them and their caregivers how to use the system on a daily basis for applications that the individual patients desire, such as e-mail, environmental control, computer-mediated conversations, word-processing, and/or entertainment. The VA teams will provide long-distance Internet-based oversight as the patients begin to use BCI technology for communication and control in their daily lives. The Project teams will be available for onsite supervision at the beginning of BCI use and for periodic in-home evaluations later on. In addition to providing ongoing oversight and guidance of the project, the group will focus on reducing the need for continued expert support (both onsite and remote) by incorporating into the BCI software adaptations and adjustments that are essential for reliable operation and by further simplifying and streamlining the caregiver interface and other aspects of system operation. The ultimate goal is a practical system that can be used by many severely disabled people in their homes with minimal ongoing technical support.

Aim 2: To assess the extent and success of BCI usage and its impact on quality of life. Via the Internet link and periodic visits, the Project teams will quantify the amount of BCI usage in both absolute terms and in terms of its importance for supporting specific functions (e.g., interactions with family, e-mail); and will quantify BCI performance in terms of accuracy and speed. In addition, standard and specialized quality-of-life measures and BCI assessment questionnaires will be used to quantitatively evaluate the long-term impact of BCI technology on the lives of the users, their caregivers, and their families. The effects of disease progression (e.g., loss of remaining neuromuscular function) on the extent and nature of BCI use will also be monitored. We expect this work to establish that the communication and control applications provided by the BCI system are heavily used by people severely disabled by ALS, that the BCI can produce lasting improvement in their lives and in the lives of those close to them, and that the BCI can even allow people who would otherwise become totally locked-in to continue to interact with their families and friends.

The success of this project will depend on establishment and maintenance of reliable high-speed daily communication between the subjects, the VA sites, and the Project team. The VA and investigators must be able to evaluate each subject's EEG data every day, 7 days/week, so that questions can be answered, problems can be solved, and system parameters can be optimized within 24 hrs.

In this study, the first primary hypothesis is that the subjects will begin to use the BCI for important purposes in their daily lives and that they will continue and even increase this use throughout the period of the study. Thus, the primary quantitative outcomes for this hypothesis will be 1) the time spent using the BCI and 2) the change in this time over the study period. If their BCI use time is substantial and remains stable or increases over the study, we will be able to conclude that the subjects have found the BCI system desirable and valuable. The second primary hypothesis is that BCI will improve the quality of life of people severely disabled by ALS. Secondary outcomes include: caregiver quality of life measures; the patient and caregiver assessments of BCI usefulness; the BCI performance (i.e., speed and accuracy); and the amount of time spent by project staff in technical support.

The completion of this study and the achievement of its aims should help to move EEG based BCI technology out of the laboratory and to demonstrate that it is a powerful, clinically practical, and affordable communication and control technology that can substantially improve the lives of people with ALS. Furthermore, the study should validate and establish an important new option, BCI-based communication that the VA can provide to many of its most severely disabled patients. This achievement would make the VA the first and only entity in the world that can provide this radically new and important assistive technology to its patients.

Forty prospective BCI Users satisfied the inclusion criteria and provided informed consent*. [*Footnote 1: Two additional people who provided informed consent were subsequently found to not satisfy the inclusion criteria.] Thirty-seven completed the BCI assessment sessions, 28 satisfied the BCI accuracy criterion, and 27 had the BCI system placed in their homes.

ELIGIBILITY:
Inclusion and Exclusion Criteria

1. Subject will be a veteran with El Escorial "Lab Supported Probable" or more definite diagnosis of ALS.
2. Subject will have lost the ability to communicate either verbally or in writing (item 1 or item 4 on the ALS Functional Rating Scale-Revised (ALSFRS-R) score of 0, Appendix A) .
3. Subject will be an adult (age >18).
4. Subject will be living at home.
5. Subject will be living within 100 miles of the participating study site.
6. Subject will have corrected visual acuity of at least 20/80.
7. Subject will have the ability to read and understand 6th grade English text on a computer screen.
8. Subject will be able to indicate willingness and understanding of the consent form (using their existing method of communication).
9. Subject will be able to identify one significant other.
10. Subject will identify one system operator (person that agrees to be trained and set up the BCI). This person can be the significant other.
11. Subject will be able to communicate non-verbally with their significant other, caregiver and system operator, and with study personnel.
12. Significant other, caregiver and system operator will be able to indicate willingness and understanding of the consent form, be adults (age> 18) and expect to be with the subject for at least one year.
13. Subject, significant other, caregiver and system operator will have life expectancy of at least one year.
14. In the opinion of the BCI installation team, the home environment is physically and technologically conducive to BCI operation and use.
15. Subject will demonstrate during the screening phase sufficient EEG interaction for the BCI to operate, i.e. classification rate of 70%. Classification rate is defined as the proportion of correct selections made during the daily calibration period of "copy spelling." Copy spelling data refers to data collected while the patient attends to and selects specific predefined characters.
16. Significant other, caregiver and system operator will demonstrate during the screening phase sufficient skill to manage the daily set-up and routine operations needed for the subject's basic operation of the BCI.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects were patients at five VA medical centers who were severely disabled by amyotrophic lateral sclerosis (ALS).
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ruff, MD PhD, Study Chair — VA Medical Center-Cleveland
Locations (5):
- United States (5):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Albany VA Medical Center Samuel S. Stratton, Albany, NY, Albany, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process was from 09/01/11 to 04/30/12. After the participants were identified they were sent a letter asking them to participate. After that screening began. The participating sites were Cleveland, Durham, West Haven, Albany, Providence.
Pre-assignment Details: Screening qualifications of baseline assessment. The participants had initial contact for interest, consent obtained, and determine electrical environment. If participant passed screening they were enrolled and had to complete training on the device.
Groups:
- BCI Device: All participants will use the BCI System as a means of communication.
  Brain Computer Interface (BCI): A Brain Computer interface or BCI records brain signals and analyzes them to derive device commands. BCIs give their users communication and control channels that do not depend on peripheral nerves and muscles.
Period: Overall Study
Arm/Group | BCI Device
Started | 27
Independent Users | 14 (All data analyses were based on the 14 independent users.)
Completed | 3
Not Completed | 24
Not completed — Death | 4
Not completed — Withdrawal by Subject | 14
Not completed — Did not complete in the timeframe | 6

BASELINE CHARACTERISTICS:
Population: Participant with ALS age more than 18, living at home within 100 miles of the pariticipating study site, visual acuity of al least 20/80, and communicate non-verbally with their significant other, caregiver and system operator, and with study personnel and demonstrate during the screening phase sufficient EEG interaction for the BCI to operate.
Arm/Group | BCI Device
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.32 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — No preference on race during recruitment.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 24
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
ALS-Functional Rating Scale-R (ALSFRS) [Mean (Standard Deviation); unit: units on a scale] — The ALS Functional Rating Scale revised includes 12 questions. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 48=best.
  units on a scale | 15 (13)

OUTCOME MEASURES:

1. Primary Outcome: BCI System Usage by the ALS Patient
Description: This study will look at the 14 independent users usage of the BCI system. The continued use will be assessed by total time.
Time Frame: Up to 18 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BCI Device
Number analyzed (Participants) | 14
days | 171 (12)

2. Secondary Outcome: BCI Usage by and Impact on the ALS Patient
Description: At three-month intervals, BCI use will be summarized. On a daily basis the BCI will record the total of number of selections made in copy spelling mode. Copy spelling mode is used for system calibration. Participants are expected to indicate that the burden associated with BCI use is inconsequential to the benefit derived from using the BCI. This will be assessed by the McGill Quality of Life (MQOL) at each visit.
Time Frame: Up to 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BCI Device: The McGill Quality of Life (MQOL) is a 16 item scale that has five distinct sub-measures: physical well-being; physical symptoms; psychological symptoms; existential well-being; support. These sub-measures are averaged to give a MQOL total score.
  The range of total score is from 0 (worst) to 10 (best).
Arm/Group | BCI Device
Number analyzed (Participants) | 14
units on a scale
  Visit 4.0 (3 month) | 6.59 (1.94)
  Visit 5.0 (6 month) | 7.75 (0.85)
  Visit 6.0 (9 month) | 6.93 (1.63)
  Visit 7.0 (12 month) | 6.52 (1.56)
  Visit 8.0 (15 month) | 7.26 (0.61)

3. Secondary Outcome: Time of BCI Impact on the Significant Other and Systems Operator
Description: The quality of life of the significant other, caregiver and system operator will be measured using the Caregiver Burden Assessment at visits. At three month intervals, the significant other, caregiver and system operator will be asked to estimate how much time they spend on the following tasks per day in minutes: BCI System setup ( placing the electrode cap and initiating system operation), BCI System cleanup, and BCI System maintenance (removing cap).
Time Frame: Up to 18 months
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- BCI Device - Time Assisting Patient With Device: All participants will use the BCI System as a means of communication.
  Brain Computer Interface (BCI): A Brain Computer interface or BCI records brain signals and analyzes them to derive device commands. BCIs give their users communication and control channels that do not depend on peripheral nerves and muscles. The time was measured of how long the the caregiver assisted the patient with the device.
Arm/Group | BCI Device - Time Assisting Patient With Device
Number analyzed (Participants) | 14
minutes
  BCI System setup | 13 (6)
  BCI System cleanup | 15 (9)
  BCI System maintenance | 4 (6)

4. Secondary Outcome: Facility Support Speed of Solution
Description: This study will look at how the technical problems of the BCI are supported by the facility through analyzing the speed of solution.
Time Frame: Up to 18 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BCI Device
Number analyzed (Participants) | 14
hours | 62 (90)

5. Primary Outcome: BCI System Usage by the ALS Patient
Description: This study will look at the 14 independent users usage of the BCI system. The continued use will be assessed by time per application.
Time Frame: Up to 18 months
Measure: Median (Standard Deviation); unit: percentage of BCI time
Arm/Group | BCI Device
Number analyzed (Participants) | 14
percentage of BCI time | 63 (20)

6. Primary Outcome: BCI System Usage by the ALS Patient
Description: This study will look at the 14 independent users usage of the BCI system. The continued use will be assessed by accuracy. Accuracy rate - The proportion of correct selections made during the daily calibration period of "copy spelling." Copy spelling data refers to data collected while the patient attends to and selects specific predefined characters, this allows the data to be coded properly (e.g., THE QUICK BROWN FOX JUMPS OVER THE LAZY DOG). Copy spelling data is used for calibration and will be collected at least 2x/week, and may be collected more frequently if unstable performance could be improved by more frequent calibration runs. The independent-use periods of the 14 independent users was totaled by days. Of these days, BCI use was not possible for days (i.e. hiatus days) due to hospitalization, illness, home construction, travel, or BCI system assistant (SA) absence. Over these days, copy-spelling accuracy was averaged.
Time Frame: Up to 18 months
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | BCI Device
Number analyzed (Participants) | 14
percentage of days | 71 (11)

7. Primary Outcome: BCI System Usage by the ALS Patient
Description: This study will look at the 14 independent users usage of the BCI system. The continued use will be assessed by selection rate. Accuracy rate - The proportion of correct selections made during the daily calibration period of "copy spelling." Copy spelling data refers to data collected while the patient attends to and selects specific predefined characters, this allows the data to be coded properly (e.g, THE QUICK BROWN FOX JUMPS OVER THE LAZY DOG). Copy spelling data is used for calibration and will be collected at least 2x/week, and may be collected more frequently if unstable performance could be improved by more frequent calibration runs. The number of selections/min for the BCI applications was averaged across users.
Time Frame: Up to 18 months
Measure: Mean (Standard Deviation); unit: number of selection per minute
Arm/Group | BCI Device
Number analyzed (Participants) | 14
number of selection per minute | 2.9 (1.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Screening until 3 months past the last follow-up visit. The period of collection 1 year and 10 months.
Description: An adverse events (AE) can be any unfavorable or unintended sign, or symptom associated with the use of the device, including psychological signs or symptoms.
  Examples of adverse events may include one of the following:An effect of the investigational product and An accident or injury related to the device
Arm/Group | BCI Device
Serious Adverse Events (participants affected / at risk) | 12/27
Other Adverse Events (participants affected / at risk) | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCI Device (N=27)
Pneumonia (Infections and infestations) | 3 (3)
Medical device complication and disease progression. (General disorders) | 2 (2)
Fall or overdose (Injury, poisoning and procedural complications) | 2 (2)
Gastrointestinal tube insertion (Surgical and medical procedures) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Respite care (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCI Device (N=27)
Fall or procedural complications (Injury, poisoning and procedural complications) | 2 (3)
Therapy cessation and gastrointestinal tube insertion (Surgical and medical procedures) | 2 (2)
Unevaluable event (General disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Some limitations would be the Caregivers willingness and ability to support BCI user. In addition, the caregivers limited availability and the time commitment of the usage of the BCI system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No